CLINICAL TRIAL: NCT06918652
Title: Surgical vs Endoscopic Treatments as ImmunoModulating Interventions in High-Risk Acute Calculous Cholecystitis
Acronym: SETIMIHRACC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Luca Ansaloni, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SETIMIHRACC
Record Dates: First submitted 2025-03-22; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: High-risk Patients With Acute Calculous Cholecystitis (ACC)
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transmural ultrasound-guided gallbladder drainage (Experimental): Patients randomized to TUGD arm will receive endoscopic transmural ultrasound-guided gallbladder drainage with lumen-apposing self-expandable metal stents (LAMSs)
  Interventions: Procedure: Transmural ultrasound-guided gallbladder drainage
- Laparoscopic cholecystectomy (Active Comparator): Patients randomized to control arm (LC) will receive laparoscopic cholecystectomy.
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Transmural ultrasound-guided gallbladder drainage — TUGD will be performed using the bi-flanged LAMSs mounted on an electrocautery-enhanced delivery system (Hot-AXIOS™) by an experienced endoscopist defined as > 10 LAMS positioning per year. The diameter and length of the stent and the modality of placing the stent (under complete EUS view or with endoscopic or fluoroscopic guidance) will be chosen at the discretion of the endoscopist performing the procedure
  Arms: Transmural ultrasound-guided gallbladder drainage
Procedure: Laparoscopic cholecystectomy — LC will be performed by the four-trocar technique with transection of the cystic duct and cystic artery after reaching the critical view of safety. ELC will be performed by a surgeon trained and experienced in laparoscopic surgery defined as > 5 laparoscopic procedures for ACC on a yearly basis
  Arms: Laparoscopic cholecystectomy

SUMMARY:
Randomized controlled trial on high-risk patients with ACC. Consecutive patients with a diagnosis of ACC, if they meet the inclusion and exclusion criteria, will be randomized to receive Laparoscopic cholecystectomy (LC) or transmural ultrasound-guided gallbladder drainage (TUGD) with lumen-apposing self-expandable metal stents (LAMSs) within 10 days from onset of symptoms. Blood cultures will be performed at the time of admission, just before the procedure, 24 ± 3h after procedure, 72 ± 3h after procedure. Bile samples will be taken during the procedure for microbiological exam and culture. Blood samples will collected from all patients at the time of admission, just before the procedure, 24 ± 3h after procedure, 72 ± 3h after procedure.

The follow-up will be performed after 30 days and after 6 months from intervention with an outpatient medical examination.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of ACC as defined by 2018 Tokyo Guidelines criteria
* be ≥ 18 years old
* have a POSSUM PS ≥ 25
* onset of symptoms <= 7 days before Emergency Department (ED) admission
* provide signed and dated informed consent form
* willing to comply with all study procedures and be available for the duration of the study
* have an Israelian Score (IS) (Table 3) for the risk of main bile duct stones <2 or an IS =2 and an EUS or a MRCP negative for main bile duct stones

Exclusion Criteria:

* Pregnancy
* Patients unwilling to undergo follow-up assessments
* Patients diagnosed with concomitant pancreatitis
* Acute cholecystitis not related to a gallstone etiology
* Onset of symptoms >7 days before ED admission
* Altered anatomy of the upper gastrointestinal tract due to surgery of the esophagus, stomach and duodenum
* Previous drainage of the gallbladder
* Biliary peritonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is to find if TUGD with LAMSs, compared to LC, has a lower inflammatory and immunologic impact on high-risk patients with ACC. | baseline, pre-surgery, day 3
  Difference between the plasma elastase concentration before surgery and on the third postoperative day

SECONDARY OUTCOMES:
difference between the plasma concentration biochemical and immunological parameters | baseline, pre-surgery, day 1, day 3
  PTX (pentraxin-1, PCR), PTX2, PTX3, SAA (serum amyloid A) , PCT (procalcitonine), C3b, Pro-adrenomedullina, Cortisol, Hepcidin, TNFalpha, IL-1, IL-6, IL-8, IL-10 and IFNgamma, total WBC count, WBC subpopulation (neutrophils and total lymphocytes), T-helper lymphocytes (CD4), T-suppressor lymphocytes (CD8), natural killer lymphocytes (CD16 and CD56), pan B cell antigen (CD20), T-cell receptor gamma/delta, T reg, Th 17, human leukocyte antigen-DR (HLA-DR)
30-day postoperative complication rate according to Clavien-Dindo | day 30
  Rate of: biliary tree injury, hemorrhage, wound infection, deep infection (collections, abscesses), urinary tract infection, bowel perforation, biliary leakage, paralytic ileus, respiratory complication, cardiac complication, renal complication, cerebrovascular complication, thrombo-embolic complication, other
30-day postoperative biliary complication rate | day 30
  Rate of biliary leakage and main biliary duct injury
30-day postoperative mortality rate | day 30
  Mortality rate
Intraoperative complication rate | day 0
  Rate of bleeding >500ml, Biliary tree injury, Bowel perforation, Major vascular injury, Anesthesia respiratory complications, Anesthesia cardiac complications, Other
Failure rate of performing the procedure | day 0
  Rate of failure
Operative times | through study completion, an average of 2 years
  * Procedure duration (measured from skin incision to skin closure for LC and from the introduction of the endoscope to its extraction for if TUGD with LAMSs) (minutes)
  * Time of occupation of the operating room (minutes)
  * Time from admission to the ED to the procedure (days)
  * rate of patients who used the prescribed painkiller "to need"
  * average of daily administrations of painkillers prescribed "to need" in the first post-procedure day
  * rate of patients where postoperative pain management therapy had to be varied compared to protocol
Postoperative length of stay (PO-LOS) | through study completion, an average of 2 years
  Postoperative length of stay (days)
Total length of stay (T-LOS) | through study completion, an average of 2 years
  Total length of stay (days)
Total readmission rate within 6 months | 6 Months after procedure
  Readmission rate for all causes
Readmission rate within 6 months due to Gallstones Relates Events (GRE) | 6 Months after procedure
  Readmission rate due to biliary colic, acute cholecystitis, acute pancreatitis, obstructive jaundice and cholangitis
Outcomes of blood and bile cultures (to define the infectious state of the patient) | Baseline, pre-surgery, during the surgery, day 1, day 3
  Outcomes of blood and bile cultures
Post-operative pain | through study completion, an average of 2 years
  rate of patients who used the prescribed painkiller "to need"
  * average of daily administrations of painkillers prescribed "to need" in the first post-procedure day
  * rate of patients where postoperative pain management therapy had to be varied compared to protocol

CONTACTS AND LOCATIONS:
Overall Officials: Luca Ansaloni, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia
Locations (1):
- SC Chirurgia Generale 1 - Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No